CLINICAL TRIAL: NCT05635435
Title: Preoperative Immune and Inflammatory Indices in Peripheral Blood Predict Prognosis of Glioma and Correlate With Grades and Subtypes: A Prospective Multi-Institutional Study
Brief Title: Immune and Inflammatory Indices in Peripheral Blood Predict Prognosis of Glioma and Correlate With Grades and Subtypes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonggao Mou, Clinical Professor, Sun Yat-sen University
Other Study IDs: ShengZhong
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Glioma; Immune Suppression
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primary glioma patients: We collected the information of clinical characteristics, inflammatory factors and immune factors of patients with primary glioma.
  Interventions: Other: Detection of Immune and Inflammatory Indices in Peripheral Blood

INTERVENTIONS:
Other: Detection of Immune and Inflammatory Indices in Peripheral Blood — We detected immune and inflammatory indices in peripheral blood at each patient's at first hospitalizatin from October 13th, 2006, to April 6th, 2022.

SUMMARY:
Our study considered the relevant immune and inflammatory indices, such as immunoglobulin kappa light chain, TNF, and CD4+ Helper T lymphocyte% in a multi-institutional study with a large patient cohort (n=1282) from the east, northeast, and southeast of China. Our study shed light on the association of peripheral immune system status with prognosis, tumor grade, and subtype of glioma, which can potentially benefit future diagnostic and prognostic processes of glioma given its noninvasive nature. Moreover, the preoperative inflammatory status can be leveraged for timely interventions to reverse the immunosuppressive status of cancer patients and enhance anti-tumour immunity of glioma.

ELIGIBILITY:
Inclusion Criteria:

* glioma grading and classification histologically verified in a resection or biopsy specimen according to 2016 WHO criteria;
* age > 18 years;
* primary malignant glioma;
* the duration of follow-up > 3 months;
* available data of lymphocyte subsets, cytokines, immune proteins and immune complements measured at the patient's first hospitalization.

Exculsion Criteria:

* current infectious disease, hyperpyrexia, hematological disease, diabetes mellitus, serious heart disease, hypertension, metabolic syndrome, severe renal or hepatic dysfunction, other cancer, autoimmune disease, inflammatory disease, or medication usage related to an inflammatory condition;
* prior cancer-specific pretreatment, such as chemotherapy or radiotherapy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In our cohort, there were more males (count, 761, percentage, 59.39%) than females. In addition, 762 patients (percentage, 59.4%) were diagnosed as grade IV glioma according to 2021 WHO criteria, which was far more than the other grades in our study. Similar characteristics were observed in the glioma subtype. IDH1 mutation status, 1p/19q codeletion status and MGMT promoter methylation status were known in 924, 771, and 855 patients, respectively. Among them, 630 of 924 patients were IDH1 mutant type, 124 of 771 patients had 1p/19q codeletion, and 369 of 855 patients were MGMT methylated. In addition, 916 patients received chemotherapy within one month after the resection of primary glioma, while 940 patients received radiotherapy postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 1282 (Estimated)
Dates: Start 2006-10-13 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 16 years
  For this study, the endpoint was all-cause mortality. Time zero was set at the time of resection of the primary tumor.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong
  - The First Bethune Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: Undecided